CLINICAL TRIAL: NCT03158714
Title: The Alabama Healthy Marriage and Relationship Education Initiative
Brief Title: Alabama Community Healthy Marriage Initiative Evaluation Project for Couples
Acronym: AHMREI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Mathematica Policy Research, Inc. (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Francesca Adler-Baeder, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-248 EP 1608
Record Dates: First submitted 2017-05-05; First posted 2017-05-18 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Marriage; Healthy Relationship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Couples Connecting Mindfully Curriculum (Experimental): Receives the Couples Connecting Mindfully curriculum over a 6 week period.
  Interventions: Behavioral: Couples Connecting Mindfully
- ELEVATE Curriculum (Experimental): Receives the ELEVATE curriculum over a 6 week period.
  Interventions: Behavioral: ELEVATE
- Control (No Intervention): No programming is offered.

INTERVENTIONS:
Behavioral: Couples Connecting Mindfully
  Other Names: CCM
  Arms: Couples Connecting Mindfully Curriculum
Behavioral: ELEVATE
  Arms: ELEVATE Curriculum

SUMMARY:
The Alabama Healthy Marriage and Relationship Education Initiative (AHMREI), a large-scale partnership among Auburn University and 9 additional implementation partners at Family Resource Centers, implements multiple program activities that respond to family needs and integrate comprehensive services to promote healthy marriages and relationships, as authorized by the Claims Resolution Act of 2010 (Pub. L. 111-291). The purpose of this study is to evaluate the efficacy of two selected couples education curricula- Elevate and Couples Connecting Mindfully. The programs are intended to improve the well-being of individuals, couples, and families in domains such as couple well-being, parenting skills, individual skills, and economic stability.

DETAILED DESCRIPTION:
In 2015, Congress provided funding for grants to provide healthy marriage and relationship services to help interested couples enhance or improve adult and family relationships. The Administration for Children and Families (ACF), within the Department of Health and Human Services (HHS), oversees these grants and provides supports to assist grantees in meeting their goals and objectives. To learn about the implementation and effects of these programs, Dr. Francesca Adler-Baeder at Auburn University was awarded a contract to conduct a local impact evaluation study. The evaluation includes impact and process studies for couples education curricula.

Couples who are eligible for the programs and agree to be in the study are randomly assigned to either one of two program groups (Elevate or Couples Connecting Mindfully) or a no-program control group. Program group members are offered program services; control group members are not offered those services. The impact study will examine whether the programs improve outcomes for individuals in couples and the children of the participants in the program group compared to outcomes of those in the control group. Members of both program and control groups are surveyed five times over 2 years: before they are randomly assigned, immediately after the curricula have been implemented (approximately 8 weeks later), and 6 months, 1 year, and 2 years after baseline. All surveys are administered via an online survey system, Qualtrics. The survey covers a range of questions related to couple relationships and interactions, individual functioning, parent-child interactions, co-parenting quality, and economic stability. The process aspect of the study will examine multiple aspects of the implementation and operation of the programs. Specifically, program attendance or dose, participant characteristics, facilitator-participant relationship, attitudes towards the program, and mechanisms of change will be considered in the process evaluation. Information for the process evaluation is obtained through the respondents' online surveys and facilitator/educator surveys.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the AHRMEI Couples Evaluation Project, the applicant must be part of a couple (as defined by the couple) in which both couple members are applying to the program and that: both members of the couple are 19 years of age or older, both members of the couple can attend the majority of the class offerings.

Exclusion Criteria:

* Does not meet the inclusion criteria.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1858 (Actual)
Dates: Start 2016-08-11 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Adler-Baeder, Ph.D., Principal Investigator — Auburn University
Locations (10):
- United States (10):
  - Auburn University, Auburn, Alabama
  - Hope Place Family Resource Center, Brewton, Alabama
  - Parents and Children Together, Decatur, Alabama
  - The Family Success Center of Etowah County, Gadsden, Alabama
  - Family Guidance Center, Montgomery, Alabama
  - Sylacauga Alliance for Family Enhancement, Sylacauga, Alabama
  - Tuscaloosa's ONE Place, Tuscaloosa, Alabama
  - Circle of Care Center for Families, Valley, Alabama
  - IMPACT Family Counseling, Vestavia Hills, Alabama
  - Alabama Cooperative Extension Syestem- Elmore County, Wetumpka, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funk JL, Rogge RD. Testing the ruler with item response theory: increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. J Fam Psychol. 2007 Dec;21(4):572-83. doi: 10.1037/0893-3200.21.4.572. PMID 18179329
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042

RESULTS

PARTICIPANT FLOW:
Groups:
- Couples Connecting Mindfully Curriculum: Receives the Couples Connecting Mindfully curriculum over a 6 week period.
  Couples Connecting Mindfully
- ELEVATE Curriculum: Receives the ELEVATE curriculum over a 6 week period.
  ELEVATE
Period: Overall Study
Arm/Group | Couples Connecting Mindfully Curriculum | ELEVATE Curriculum | Control
Started | 626 (Number of participants enrolled and Started represents number of individual participants rather than couples) | 626 (Number of participants enrolled and Started represents number of individual participants rather than couples) | 606 (Number of participants enrolled and Started represents number of individual participants rather than couples)
Completed | 445 (Participated in half or more of program.) | 398 (Participated in half or more of program.) | 606 (All control group participants completed the control protocol (no program).)
Not Completed | 181 | 228 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Couples Connecting Mindfully Curriculum | ELEVATE Curriculum | Control | Total
Number analyzed (Participants) | 626 | 626 | 606 | 1858
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Some participants did not fill out complete age information on the baseline survey, so we are missing this demographic data on a few participants for each group (ELEVATE, CCM, and Control)
  Years
    number analyzed (Participants) | 607 | 607 | 584 | 1798
    (all) | 38.17 (12.85) | 37.23 (11.70) | 36.46 (11.19) | 37.30 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312 | 316 | 308 | 936
  Male | 314 | 310 | 298 | 922
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 36 | 31 | 97
  Not Hispanic or Latino | 573 | 568 | 550 | 1691
  Unknown or Not Reported | 23 | 22 | 25 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 1 | 8
  Asian | 7 | 6 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 212 | 201 | 207 | 620
  White | 364 | 372 | 351 | 1087
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 38 | 45 | 42 | 125
Education Level [Count of Participants; unit: Participants]
  No degree or diploma earned | 33 | 36 | 33 | 102
  General Education Development (GED) | 48 | 55 | 39 | 142
  High School Diploma | 70 | 84 | 83 | 237
  Vocational/Technical Certification | 29 | 17 | 23 | 69
  Some college but no degree completion | 142 | 117 | 108 | 367
  Associate's Degree | 52 | 53 | 49 | 154
  Bachelor's Degree | 129 | 126 | 142 | 397
  Advanced Degree | 103 | 116 | 106 | 325
  Not Reported | 20 | 22 | 23 | 65
Relationship Status [Count of Participants; unit: Participants]
  Committed (not engaged/married) | 131 | 119 | 137 | 387
  Engaged to be married | 50 | 45 | 66 | 161
  Married | 413 | 424 | 376 | 1213
  Separated | 6 | 5 | 0 | 11
  Not Reported | 26 | 33 | 27 | 86
Parent Status [Count of Participants; unit: Participants]
  Parent | 431 | 432 | 428 | 1291
  Not a parent | 164 | 167 | 140 | 471
  Not reported | 31 | 27 | 38 | 96

OUTCOME MEASURES:

1. Primary Outcome: Couple Satisfaction Index
Description: Couple satisfaction was measured using an abbreviated version of the Couple Satisfaction Index utilized in previously published studies. The 3 items (rated from 1 [Not at all] to 6 [Completely]) are: "I have a warm and comfortable relationship with my partner," "How rewarding is your relationship with your partner?" and "In general, how satisfied are you with your relationship?" Mean composites were calculated, and the total scale ranges from 1 to 6. Higher scores indicate higher couple satisfaction.
Time Frame: 6 months
Population: 406 ELEVATE respondents, 432 CCM respondents, and 426 Control respondents completed baseline, immediate follow-up, and 6-month follow-up surveys and completed all of the CSI items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Couples Connecting Mindfully Curriculum | ELEVATE Curriculum | Control
Number analyzed (Participants) | 432 | 406 | 426
score on a scale | 4.82 (1.11) | 4.90 (1.17) | 4.78 (1.16)
Statistical Analysis 1: Comparison: ELEVATE Curriculum vs Control; Test type: Superiority; p = .005, Mixed Models Analysis — The a priori threshold for statistical significance was .05; Utilized multi-level modeling to account for nested data (individuals within couples), and accounted for time within individual; Mean Difference (Net) = .033
Statistical Analysis 2: Comparison: Couples Connecting Mindfully Curriculum vs Control; Test type: Superiority; p = .101, Mixed Models Analysis — The a priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = .020

2. Primary Outcome: The Couple Relationship Skills Inventory
Description: Couple relationship skills were measured using 32 items from the Couple Relationship Skills Inventory (CRSI). This measure was constructed to match the core relationship skills and predictors of couple quality emphasized in the HMRE programs provided. Items were taken from established and validated social science measures assessing commitment, intimate partner knowledge, friendship, caring behaviors, conflict management, and external support. Example items include, "I commit effort every day to making my relationship work," "I know my partner's current life stresses," "When things 'get heated' I suggest we take a break to calm down," and "I initiate physical affection with my partner." Items ranged from 1 (Very strongly disagree) to 7 (Very strongly agree). Composite sum scores were created at the individual level and the total scale ranges from 1-224 (i.e., 32*7 = 224). Higher scores indicate greater couple relationship skills.
Time Frame: 8 weeks
Population: 497 ELEVATE respondents, 520 CCM respondents, and 521 Control respondents completed both baseline & immediate follow-up surveys, as well as 80% of the CRSI items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Couples Connecting Mindfully Curriculum | ELEVATE Curriculum | Control
Number analyzed (Participants) | 520 | 497 | 521
score on a scale | 171.14 (24.23) | 170.73 (24.33) | 167.64 (22.85)
Statistical Analysis 1: Comparison: ELEVATE Curriculum vs Control; Test type: Superiority; p < .001, Regression, Linear — The a priori threshold for statistical significance was .05; Utilized multi-level modeling to account for nested data (individuals within couples), and controlled for baseline levels of outcome in regression; Mean Difference (Net) = 3.96
Statistical Analysis 2: Comparison: Couples Connecting Mindfully Curriculum vs Control; Test type: Superiority; p < .001, Regression, Linear — The a priori threshold for statistical significance was .05; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = 4.09

3. Primary Outcome: Individual Mental Health
Description: Individual mental health was measured using the SF-12 Mental Component Summary score assessing anxiety, depression, sense of wellbeing, and social/emotional functioning. Per the measure's design, items were asked on differing scales (e.g., 1 to 3 or 1 to 5) with different anchor responses (e.g., all of the time to none of the time, or not at all to extremely). Example items include, "During the past month how much of the time have you accomplished less than you would like" or "During the past month how often have you felt downhearted and depressed?" The SF-12 Mental Component Summary score has shown scale reliability and validity in empirical studies. Scores range from 0 to 100 with a mean of 50 and SD of 10 in the general U.S. population. Higher scores indicate better individual mental health.
Time Frame: 6 months
Population: 389 ELEVATE participants, 423 CCM participants, and 416 control respondents completed baseline, immediate post-program, and 6-month follow-up surveys, as well as 100% of the items of the SF-12 measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Couples Connecting Mindfully Curriculum | ELEVATE Curriculum | Control
Number analyzed (Participants) | 423 | 389 | 416
score on a scale | 43.63 (10.16) | 43.16 (10.28) | 43.95 (10.32)
Statistical Analysis 1: Comparison: ELEVATE Curriculum vs Control; Test type: Superiority; p = .003, Mixed Models Analysis — The a priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = .343
Statistical Analysis 2: Comparison: Couples Connecting Mindfully Curriculum vs Control; Test type: Superiority; p = .152, Mixed Models Analysis — The a priori threshold for statistical significance was .05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = .172

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed because the program in the current study is educational in nature and there were no risk of adverse events or mortality.
Arm/Group | Couples Connecting Mindfully Curriculum | ELEVATE Curriculum | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Measures were limited to self-report, which represent the participant's subjective perspective of skills and individual/relationship functioning.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT03158714/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT03158714/ICF_001.pdf